CLINICAL TRIAL: NCT03147001
Title: Nutritional Strategies for Optimizing Adaptations and Recovery Following Training 'Low'.
Brief Title: Protein Ingestion Before Training Low
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Foods (Industry); Team Denmark (Other); Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Mette Hansen, Assistant professor, PhD, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 50968
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Protein Metabolism
Keywords: Endurance exercise; Dietary protein

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking was done by providing similar tasting drinks at both trails. One was placebo, one was protein a drink
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein ingestion (Experimental): Subjects ingested protein drinks
  Interventions: Other: Protein ingestion
- Placebo (Placebo Comparator): Subjects ingested a non-caloric placebo drink
  Interventions: Other: Non-caloric placebo ingestion

INTERVENTIONS:
Other: Protein ingestion — A protein drink was ingested prior to the 90min bike ride in one of the completed trails (order randomised).
  Arms: Protein ingestion
Other: Non-caloric placebo ingestion — A placebo drink was ingested prior to the 90min bike ride in one of the completed trails (order randomised).
  Arms: Placebo

SUMMARY:
A randomized interventions study using a crossover design. Ten well trained triathletes or bikeriders will be included for to undergo two trail separated by about 3 weeks. The night before the trail each subject will performe a high intense interval trainings session on an ergometer bike. during the night an infusion of aminoacid tracers will be initiated. The subject is woken at 6.30 a.m. Blood samples and a musclebiopsy will be collected prior to the morning bike ride at 8.00a.m. Immediately before the morning bike ride is started the subject will ingest a drink of 0,5g protein or a non-caloric placebo (random order). During the bike ride and the following 4,5 hours blood will be drawn with regular intervals. at time point 0, 60 and 180 min after the training session biopsies are collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy well-trained triathletes or cyclists
* VO2max > 55 ml O2/kg/min
* Training and has been training more than 7 times a week the last 6 months.

Exclusion Criteria:

* VO2max < 55 ml O2/kg/min
* Has chronic disease
* has incjected with tracer on a previous occasion.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Muscle protein fractional synthetic rate (FSR) | FSR was measure over at time period of six hours

SECONDARY OUTCOMES:
Tracer kinetics dilution model | six hours
  A-V tracer dilution model was applied across the forearm.
Muscle signalling | Determined in biopsies sampled before and immediatly after 90min exercise in addition to one and four hours after exercise.
  Muscle signalling will be determined using western blotting in each muscle biopsy
Nitrogen excretion | Urine is collected during two periods. Collection period one: 12 hours prior to morning exercise. Collection period 2: During and four hours following exercise. Blood samples is drawn repeatedly from before to four hours after exercise.
  nitrogen excretion is determined by Plasma and urinary carbide analysis as well as plasma NH4+.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen MS, Holm L, Svart MV, Hjelholt AJ, Bengtsen MB, Dollerup OL, Dalgaard LB, Vendelbo MH, van Hall G, Moller N, Mikkelsen UR, Hansen M. Effects of protein intake prior to carbohydrate-restricted endurance exercise: a randomized crossover trial. J Int Soc Sports Nutr. 2020 Jan 28;17(1):7. doi: 10.1186/s12970-020-0338-z. PMID 31992300